CLINICAL TRIAL: NCT00956202
Title: Immunogenicity and Safety of Multiple Formulations of an Intramuscular Inactivated, Split Virion Swine-Origin A/H1N1 Influenza Vaccine With and Without Adjuvant in Healthy European Subjects Aged 3 to 17 Years
Brief Title: A Study of Inactivated Swine-Origin A/H1N1 Influenza Vaccines in Healthy European Subjects Aged 3 to 17 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GPF08; UTN: U1111-1111-4962 (Other: WHO); 2009-013346-83 (EudraCT Number)
Record Dates: First submitted 2009-08-03; First posted 2009-08-11 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Influenza; Swine-origin A/H1N1 Influenza
Keywords: Influenza; Pandemic Flu; Swine-origin A/H1N1 Influenza; Inactivated split-virion vaccine; Adjuvant
MeSH Terms: conditions — Influenza, Human | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A/H1N1 Vaccine Group 1 (Experimental): All participants will receive A/H1N1 Influenza vaccine formulation 1 at Visits 1 and 2; a subset will receive a trivalent influenza vaccine (TIV) at Month 13 (antibody persistence subset).
  Interventions: Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated)
- A/H1N1 Vaccine Group 2 (Experimental): All participants will receive A/H1N1 Influenza vaccine formulation 2 at Visits 1 and 2; a subset will receive a trivalent influenza vaccine (TIV) at Month 13 (antibody persistence subset).
  Interventions: Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated + Adjuvant)
- A/H1N1 Vaccine Group 3 (Experimental): Participants will receive A/H1N1 Influenza vaccine formulation 3
  Interventions: Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated + Adjuvant)

INTERVENTIONS:
Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated) — 0.5 mL, Intramuscular on Day 0 and Day 21 (all participants); and 0.5 mL of a trivalent influenza vaccine (TIV) at Month 13 (antibody persistence subset)
  Arms: A/H1N1 Vaccine Group 1
Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated + Adjuvant) — 0.5 mL, Intramuscular on Day 0 and Day 21 (all participants); and 0.5 mL of a trivalent influenza vaccine (TIV) at Month 13 (antibody persistence subset).
  Arms: A/H1N1 Vaccine Group 2
Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated + Adjuvant) — 0.5 mL, Intramuscular on Day 0 and day 21
  Arms: A/H1N1 Vaccine Group 3

SUMMARY:
The purpose of this study is to generate data on immunogenicity and safety of the monovalent H1N1 vaccine in support of the development and registration.

Primary objectives:

* To describe the immune response to vaccines 21 days after each vaccination in all participants.
* To describe the antibody persistence eight months after the first vaccine administration using HAI method, in a subset of participants who received two injections.
* To describe the immune response against the A/H1N1 strain using HAI method 21 days after a vaccination with the 2010-2011 NH seasonal TIV administered approximately 13 months after the first vaccination in the subset of participants who received two injections.
* To describe the safety profile of each vaccine in all participants.

DETAILED DESCRIPTION:
All participants will receive two injections of their randomized vaccine on Day 0 and Day 21, respectively.

A subset of children and adolescents participants eligible for the antibody persistence evaluation were sampled 8 months after the first vaccination, they will also be proposed to receive the 2010-2011 Northern Hemisphere (NH) seasonal Trivalent Influenza Vaccine (TIV) 13 months after the first vaccination. Immunogenicity response will be evaluated before vaccination and 21 days after vaccination with TIV, respectively.

ELIGIBILITY:
Inclusion Criteria :

All subjects:

* Provision of Informed Consent Form signed by the subject's parent(s)/legal representative (and by an independent witness if required by local regulations). In addition, provision of Assent Form signed by subjects aged 8 to 12 years, and of Informed Consent Form signed by subjects >12 years.
* Subject and parent/guardian are able to attend all scheduled visits and to comply with all trial procedures

Subjects aged 12 to 17 years:

* Aged 12 to 17 years on the day of inclusion
* For a female of childbearing potential, use of an effective method of contraception or abstinence for at least 4 weeks prior to the first vaccination, until at least 4 weeks after the last vaccination.

Subjects aged 3 to 11 years:

* Aged 3 to 11 years on the day of inclusion

At Visit 05 (Month 8), for antibody persistence assessment:

* Having received two injections of the 15 µg HA vaccine (Group 1) or of the 3.8 µg HA + AF03 vaccine (Group 2)
* Addendum 1 to Informed Consent Form has been signed by the subject's parent(s)/guardian(s) (and by an independent witness if required by local regulations). In addition, provision of addendum 1 to Assent Form signed by subjects aged 6 to 11 years, and of addendum 1 to Informed Consent Form signed by subjects ≥ 12 years.

At Visit 06, for participants eligible for the Antibody persistence evaluation who will receive the 2010-2011 Northern Hemisphere (NH) seasonal Trivalent Influenza Vaccine:

* Addendum 2 to Informed Consent Form has been signed by the subject and/or subject's parent(s)/guardian(s) (and by an independent witness if required by local regulations). In addition, provision of addendum 2 to Assent Form signed by subjects aged 6 to 11 years, and of addendum 2 to Informed Consent Form signed by subjects ≥ 12 years.

Exclusion Criteria:

All subjects:

* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Receipt of any vaccine in the 4 weeks preceding the trial vaccinations
* Planned receipt of any vaccine prior to the Day 42 blood sample
* Receipt of blood or blood-derived products in the past 3 months which might interfere with the assessment of immune response
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B antigen, or Hepatitis C as reported by parents/legal representative
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances
* Thrombocytopenia contraindicating intramuscular (IM) vaccination as reported by parents/legal representative
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion contraindicating IM vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Chronic illness that in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Employee of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members of the employees or the Investigator
* Previous participation in a trial investigating a vaccine with the swine-origin A/H1N1 influenza strain
* Confirmed infection with the swine-origin A/H1N1 influenza strain (different from the seasonal strain) in 2009
* Febrile illness (temperature ≥38.0°C) or moderate or severe acute illness/infection on the day of vaccination, according to Investigator judgment
* Receipt of any allergy shots and/or seasonal allergy medication in the 7-day period prior to enrollment (vaccination), or scheduled to receive any allergy shots and/or seasonal allergy medication in the 7-day period after enrollment (vaccination)

Subjects aged 12 to 17 years:

* Known pregnancy, or a positive urine pregnancy test
* Currently breastfeeding a child
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures

At Visit 05 (Month 8), for antibody persistence assessment:

* Subjects who received, in the context of a pandemic immunization program, another A/H1N1 pandemic influenza vaccine than the Investigational Medicinal Products.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 303 (Actual)
Dates: Start 2009-08; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: To provide information concerning the immunogenicity of Swine A/H1N1 influenza vaccines | 21 days post vaccination
Safety: To provide information concerning the safety (in terms of solicited injection site and systemic reactions and unsolicited adverse events) of Swine A/H1N1 influenza vaccines. | 0-7 days post-vaccination and entire study duration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (13):
- Finland (13):
  - Espoo
  - Helsinki
  - Jarvenpaa
  - Kokkola
  - Kotka
  - Kuopio
  - Lahti
  - Oulu
  - Pori
  - Seinäjoki
  - Tampere
  - Turku
  - Vantaa

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com